CLINICAL TRIAL: NCT00449722
Title: Double-blind, Double-dummy, Randomised, Multicentre, Comparative Study of the Efficacy and Tolerability of Once Daily 3.0 g Mesalazine Granules Versus Three Times Daily 1.0 g Mesalazine Granules in Patients With Active Ulcerative Colitis
Brief Title: OD vs. TID Dosing With Mesalazine Granules in Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAG-26/UCA; 2004-001216-31
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mesalazine

SUMMARY:
To proof the therapeutic equivalence of once daily (OD) versus three times daily (TID) dosing of total 3.0 g mesalazine granules in patients with active ulcerative colitis

ELIGIBILITY:
Inclusion Criteria (main):

* Active ulcerative colitis except proctitis, i.e. inflammation minimal 15cm ab ano, confirmed by endoscopy and histology
* Established or new diagnosis
* Disease activity at baseline: Clinical Activity Index (CAI) >4 and Endoscopic Index (EI) >= 4

Exclusion Criteria (main):

* Crohn's disease
* Toxic megacolon
* Present or past colorectal cancer
* Symptomatic gastrointestinal disease
* Serious secondary disease(s)
* Baseline stool positive for germs causing bowel disease
* Immunosuppressants within 3 months and/or corticosteroids within 1 month prior to baseline
* Current relapse occurred under maintenance treatment with >2g/day mesalazine
* Serum creatinine >= 1.2x upper limit of normal (ULN) and creatinine clearance < 60 ml/min per 1.73 m2
* Serum transaminase (ALT and/or AST), and/or alkaline phosphatase >= 2x ULN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission

SECONDARY OUTCOMES:
Rate of clinical response
time to resolution of symptoms
rate of endoscopical remission
rate of endoscopical response
rate of histological remission
rate of histological response
PGA

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kruis, Professor, Principal Investigator — Evangelisches Krankenhaus Kalk, Cologne, Germany
Locations (1):
- Evangelisches Krankenhaus Kalk, Cologne, Germany

REFERENCES:
- [Result] Kruis W, Kiudelis G, Racz I, Gorelov IA, Pokrotnieks J, Horynski M, Batovsky M, Kykal J, Boehm S, Greinwald R, Mueller R; International Salofalk OD Study Group. Once daily versus three times daily mesalazine granules in active ulcerative colitis: a double-blind, double-dummy, randomised, non-inferiority trial. Gut. 2009 Feb;58(2):233-40. doi: 10.1136/gut.2008.154302. Epub 2008 Oct 2. PMID 18832520